CLINICAL TRIAL: NCT03387943
Title: A Prospective, Multicenter, Open Label Phase Ⅱ Clinical Trial of Doxorubicin Hydrochloride Liposome Injection Combined With Cisplatin in the Treatment of Advanced Poorly Differentiated Thyroid Carcinoma
Brief Title: PLD Combined With Cisplatin in the Treatment of Advanced Poorly Differentiated Thyroid Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-CG-01
Record Dates: First submitted 2017-12-11; First posted 2018-01-02 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-02

CONDITIONS: Poorly Differentiated Thyroid Carcinoma
MeSH Terms: interventions — 1-dodecylpyridoxal; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLD plus Cisplatin (Experimental): liposomal doxorubicin(PLD) 35 mg/m2,iv,d1, plus cisplatin 75 mg/m2,drip,d1-3, once every 21days, for 6 cycles, to progression or intolerance.
  Interventions: Drug: PLD; Drug: Cisplatin

INTERVENTIONS:
Drug: PLD — intravenous infusion of liposomal doxorubicin 35 mg/m2, d1,once every 21days, for 6 cycles.
  Other Names: duomeisu
Drug: Cisplatin — cisplatin 75 mg/m2, drip, total dose should be carried out on d1-3; once every 21days, for 6 cycles.
  Other Names: shunbo

SUMMARY:
This is a prospective, multicenter, open label Phase II Clinical Trial. 30 advanced poorly differentiated thyroid carcinoma patients who were histopathologically confirmed inoperable were enrolled in this study.

DETAILED DESCRIPTION:
Subjects will receive the treatment regimen as follow:

intravenous infusion of liposomal doxorubicin 35 mg/m2, d1; cisplatin 75 mg/m2, drip, total dose should be carried out on d1-3; once every 21days, for 6 cycles. Stop the treatment if the patients have progressed or intolerated to the toxicity. The primary endpoint is disease control rate(DCR), the secondary endpoint is overall survival (OS), progression-free survival (PFS), safety and quality of life assessment(QoL).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate and sign the informed consent form;
2. Age :18-70 years old;
3. Histopathologically confirmed inoperable advanced poorly differentiated thyroid carcinoma;
4. Previously received surgery, I131 treatment, radiotherapy, chemotherapy patients can be enrolled；
5. At least one measurable lesion according to the solid tumor efficacy evaluation criteria (RECIST 1.1);
6. Expected survival time ≥ 3 months;
7. Karnofsky score ≥70;
8. Blood test：ANC ≥1.5×109/L； PLT ≥75×109/L；Hb ≥90g/L;
9. Liver function:Serum bilirubin (SB) level:≤ normal upper limit（ULN）2 times; aspartate aminotransferase(AST) and alanine aminotransferase(ALT) ≤ ULN 2.5times; or ≤ ULN 5times if Liver metastases are present;
10. Renal function: Serum creatinine ≤ ULN 1.5times;
11. LVEF ≥ 50%;
12. No serious complications such as active digestive tract hemorrhage, perforation, jaundice, gastrointestinal obstruction, noncancerous fever > 38℃;
13. Subjects are well-behaved, able to undergo the follow-up efficacy and adverse reactions according to the program requirements.

Exclusion Criteria:

1. Active or uncontrolled severe infection (≥CTCAE grade 2 infection)；
2. Previously received anthracycline-based regimen: the cumulative dose of doxorubicin at or above 500 mg / m2 or the cumulative dose of epirubicin reached or exceeded 800 mg / m2;
3. The New York Heart Association (NYHA) graded class II or above heart disease patients previously or at present;
4. Patients with CNS disorders or CNS metastases;
5. Allergic to chemotherapeutic drugs or their excipients or intolerant patients;
6. Received any other test drug treatment within 30 days of the first chemotherapy administration;
7. Pregnant or lactating women;
8. Arterial/venous thrombosis occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis, and pulmonary embolism;
9. History of aneurysm;
10. Neurological disorders with a history of epilepsy or ataxia require treatment;
11. A history of drug abuse and incapable of abstinence or mental disorder;
12. A history of peripheral neuropathy and the muscle strength is below level 3;
13. Suffering from other diseases and complications of hand-foot syndrome;
14. Researchers think it is not suitable for enrolling.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
disease control rate(DCR) | disease control rate will be evaluated every 2 cycles (each cycle is 21 days) from date of administration of drugs until the date of first documented progression，up to 18 months.
  the rate of CR,PR and SD

SECONDARY OUTCOMES:
OS | From date of randomization until the date of death from any cause,assessed up to 18 months.
  overall survival
PFS | From date of randomization until the date of first documented disease progression or date of death from any case,whichever came first,assessed up to 18 months.
  progression-free survival
Incidence of adverse events assessed by number and severity of adverse event in the treatment. | A summary of adverse events of each cycle,from date of administration of drugs until 30 days after the last chemotherapy or progression,whichever came first,assessed up to 18 months.
  Evaluate the adverse reaction rate of drugs assessed by number and severity of adverse events in the treatment of advanced thyroid poorly differentiated carcinoma.
quality of life assessment | It will be assessed before the administration of drugs at each first day of the chemotherapy cycle,up to 6 cycles,each cycle is 21 days.
  Evaluate the QoL according to Functional Assessment of Cancer Therapy.

CONTACTS AND LOCATIONS:
Overall Officials: minghua ge, doctor, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Zhejiang, China